CLINICAL TRIAL: NCT06893354
Title: Explore the Mechanisms Underlying Disease Resistance and Potential Primary Resistance Mechanism of Induction Therapy Lorlatinib in Resectable Non-small Cell Lung Cancer (NSCLC) Harboring ALK Positive Mutation Revealed by Single-cell RNA Sequencing and Spatial Transcriptomics
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Chief physician, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LORLAL-001-V1
Record Dates: First submitted 2025-03-07; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: NSCLC
MeSH Terms: interventions — lorlatinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lorlatinib group (Experimental)
  Interventions: Drug: lorlatinib
- lorlatinib plus chemotherapy group (Active Comparator)
  Interventions: Drug: lorlatinib plus chemotherapy

INTERVENTIONS:
Drug: lorlatinib — Subjects will be registered to receive oral lorlatinib 100mg qd for 3 cycles of 4 weeks each (12 weeks total), and then underwent surgery.
  Arms: lorlatinib group
Drug: lorlatinib plus chemotherapy — Subjects will be registered to receive oral lorlatinib 100mg qd for 3 cycles of 4 weeks each (12 weeks total) plus chemotherapy, and then underwent surgery.
  Arms: lorlatinib plus chemotherapy group

SUMMARY:
This is an open-label, randomized, single-center study. This translational study aims to explore tumor microenvironment remodelling after induction therapy lorlatinib and identify mechanisms of disease persistence and potential primary resistance mechanisms of lorlatinib as induction therapy treatment in surgically resectable ALK-rearranged NSCLC by single-cell RNA sequencing (scRNA-seq) and Spatial transcriptomics.

DETAILED DESCRIPTION:
to explore tumor microenvironment remodelling after induction therapy lorlatinib and identify mechanisms of disease persistence and potential primary resistance mechanisms of lorlatinib as induction therapy treatment in surgically resectable ALK-rearranged NSCLC by single-cell RNA sequencing (scRNA-seq) and Spatial transcriptomics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are ≥18 years of age；
* Histologically or cytologically documented non-squamous NSCLC with completely resectable (Stage IB-III) disease
* Clinical stage IIA/IIB/IIIA/IIIB assessed by EBUS-TBNA or PET(positron emission tomography)/CT can be resected.
* Documented ALK-fusion positive（ Ventana , assessed by a local laboratory）
* ECOG PS 0-1
* Performance status (ECOG) 0-1 at enrolment, with no deterioration over the previous 2 weeks prior to baseline or day of first dosing of lorlatinib
* Hematology , liver and kidney function are adequate for induction therapy .
* Cardiopulmonary function suitable for surgical treatment (ECG, echocardiography, pulmonary function or blood gas analysis).
* Be willing and able to provide written informed consent for the trial prior to any study specific procedures. The subject must also provide consent for correlative translational study.
* Female participants of childbearing potential must agree to use acceptable methods of contraception
* Male patients must be willing to use barrier contraception. Provide written informed consent.

Exclusion Criteria:

* Mixed squamous cell carcinoma, large cell carcinoma, small cell lung cancer.
* Prior treatment with any systemic anti-cancer therapy for NSCLC including chemotherapy, biologic therapy, immunotherapy, or any investigational drug.
* Pregnant female patients; breastfeeding female patients.
* Malignancies other than the disease under study within 3 years prior to Cycle 1, Day 1, with the exception of patients with a negligible risk of metastasis or death and with expected curative outcome
* Severe infection within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infections, or any active infection that, in the opinion of the investigator, could impact participant safety
* Pregnant or lactating, or intending to become pregnant during the study Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Single-cell RNA sequencing (scRNA-seq) | Obtain the primary tumor tissue before drug administration; after the end of cycle 3（each cycle is 28 days) of induction therapy, the fresh tumor tissues will be collected immediately by surgical resection.
  use the Singleron Matrix® Single Cell Processing System (Singeleron) according to the manufacturer's instructions to conduct the single-cell experiment and sequencing. It will be performed by an authorized, qualified independent laboratory.

IPD SHARING:
Plan to Share IPD: No